CLINICAL TRIAL: NCT03429686
Title: The Use of Digital Technology in Reminiscence Work With People With Dementia in Jordanian Care Homes: A Feasibility Study
Brief Title: Digital Reminiscence for People With Dementia
Acronym: DTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Holly Blake, Associate Professor of Behavioural Science, Faculty of Medicine & Health Sciences, University of Nottingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110-1709
Record Dates: First submitted 2018-01-24; First posted 2018-02-12 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Dementia
Keywords: dementia; reminiscence therapy; touch screen technology; digital reminiscence therapy
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: A single group pre-post intervention feasibility study with process evaluation. Data will be collected from residents and staff in Jordanian care homes through questionnaires, from care home records, and qualitative interviews.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DRT Intervention (Experimental): Intervention: Individual digital reminiscence therapy programme.
  Interventions: Other: DRT Intervention

INTERVENTIONS:
Other: DRT Intervention — The digital reminiscence therapy intervention will run 12 sessions twice per week, for six weeks, for up to an hour at a time (this will depend on the participant's ability and willingness to participate). The sessions of reminiscence therapy will be culturally appropriate and based on the key stages in the life which most people will have experienced. These sessions are individual, face-to-face sessions.
  Other Names: Digital Reminiscence Therapy Intervention

SUMMARY:
The purpose of this study is to explore the feasibility and acceptability of a digital reminiscence therapy (DRT) intervention for people with dementia (PwD). The objectives of this study include:

1. To determine whether DTR can be delivered as planned in the care of PwD in Jordanian care homes.
2. To determine whether DTR is acceptable/tolerable to PwD and care home staff in Jordanian care homes
3. To identify the most appropriate outcome measures to evaluate the delivery of DRT to PwD in Jordanian care homes to be used in a subsequent definitive trial.

DETAILED DESCRIPTION:
Reminiscence Therapy has been shown to be beneficial for people with dementia. The aim of this research is to develop and evaluate the feasibility of a digital application to aid reminiscence for people with dementia.

This study proposes to design an application, based upon reminiscence therapy, which can act as storage for personal and communal 'positive memories' in a range of media types. This includes pictures, videos and audio.

The target for this application is people with dementia and their staff caregivers. The study aims to recruit 40-50 participants (40 PwD and 10 staff caregivers). This research will look at the requirements for developing and evaluating a mobile application to see whether it might be used to aid reminiscence for people with dementia. Additionally, this research will ensure whether this digital reminiscence therapy can be delivered and accepted as planned in the care of people with dementia in Jordanian care homes. The acceptance of this digital reminiscence therapy will be assessed by using semi-structured interviews with approximately 15 people with dementia and staff care-givers. Quantitative measures will be used before and after the intervention to explore whether certain outcomes are sensitive to change. These outcomes include memory, communication, anxiety, depression, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* People who have been clinically diagnosed with dementia determined by psychiatrist in the selected care homes. The diagnosis will be recorded in their care home notes.
* People who are residents in the designated care home and they are anticipated to be resident in the care home for the coming year.
* People who have the capacity to understand and consent to participate in the study (including those who can consent in the moment), OR they will have a consultee who can be approached for their assent if they are not able to consent in the moment but meet the eligibility criteria.

Exclusion Criteria:

* People who are deemed too unwell to participate determined by care home staff.
* People with a diagnosis of an additional psychiatric disorder other that those identified in the inclusion criteria (e.g. schizophrenia, MDD) determined by care home staff.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of the digital reminiscence therapy for PwD | 3 months
  Assessed by recruitment rate

SECONDARY OUTCOMES:
Acceptability of the digital reminiscence therapy for PwD | 3 months
  Assessed by qualitative interview data - analysis will determine participant enjoyment of the intervention, barriers to programme use, and reasons for non-adherence and attrition
Adherence to intervention | 3 months
  Assessed by adherence rate (number of sessions completed)
Study attrition | 3 months
  Assessed by % lost to attrition
Explore whether outcome measures are sensitive to change - for memory | 3 months
  Pre-post changes in Arabic Version of Saint-Louis-University-Mental-Status (SLUMS; Abdelrahman & El Gaafary, 2014) it is a 30-point, 11 questions. The maximum score is 30 points.
  Cut-off scores based on high School Education:
  21-26 = Mild Neurocognitive Impairment, 1-20 = Dementia.
  Less than High School Education:
  20-24 = Mild Neurocognitive Impairment, 1-19 = Dementia.
Explore whether outcome measures are sensitive to change - for quality of life | 3 months
  Older People's Quality of Life Questionnaire (OPQOL-brief-13; Bowling et al., 2012) Each of the 13 items is scored from 1 to 5. The items are summed for a total OPQOL-Brief, then positive items are reverse coded, so that higher scores represented higher QoL.
Explore whether outcome measures are sensitive to change - for anxiety and depression | 3 months
  Arabic version of Hospital Anxiety and Depression Scale (Arabic HADS; Al Aseri et al., 2015) it comprises 7 questions for anxiety and 7 questions for depression. each subscale is ranged from 0 to 3. Cut-off scores for both is 8 separately; 8-10: mild, 11-14: moderate, 15-21: severe.
Explore whether outcome measures are sensitive to change - for communication | 3 months
  Holden Communication Scale for Persons with Dementia (HCS; Strøm et al., 2016). it includes 12 items. each subscale is scored from 0 to 4. The total scores range from 0-48 and the higher score the more difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Blake, Dr, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No